CLINICAL TRIAL: NCT03947398
Title: A Prospective, Multi-Center Registry, Randomized Trial for Evaluation of Effectiveness of the Blimp Scoring Balloon in Lesions Not Crossable With Conventional Balloon or Microcatheter.
Brief Title: The BLIMP Balloon in Coronary Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); AZ Sint-Jan AV (Other); CHU de Charleroi (Other); Jolimont, La Louviere (Unknown); Centre Hospitalier Universitaire Saint Pierre (Other); Onze Lieve Vrouwziekenhuis Aalst (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other); University Ghent (Other); University Hospital, Antwerp (Other); Centre Hospitalier du Luxembourg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S61686
Record Dates: First submitted 2019-03-28; First posted 2019-05-13 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2019-03

CONDITIONS: Percutaneous Coronary Intervention; Chronic Total Occlusion of Coronary Artery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with BLIMP first (Experimental)
  Interventions: Device: BLIMP balloon
- Treatment with low-profile balloon first (Active Comparator)
  Interventions: Device: Low profile balloon

INTERVENTIONS:
Device: BLIMP balloon — Using BLIMP balloon to cross lesion
  Arms: Treatment with BLIMP first
Device: Low profile balloon — using low profile balloon to cross lesion
  Arms: Treatment with low-profile balloon first

SUMMARY:
The purpose of this study is to investigate the effectivness of the Blimp Scoring balloon compared to current available CTO balloon catheters.

DETAILED DESCRIPTION:
For this study two case situations are being considered.

6.1.1 Case Situation A Guidewire crossed the lesion, micro catheter does not cross

Case situation A is the circumstansis where a physician is using a guidewire in combination with a micro catheter. When in such case the guidewire is crossing at a certain moment of the procedure and the micro catheter not a balloon crossing attempt is one of the current common options as next step.

For the study the physician will go through following steps

1. select alternating in 50% of these cases his current first choice regular balloon (≤ 1.5 (mm) OD) and in the other 50% of cases the Blimp.
2. If first choice regular balloon does not cross select the Blimp and if the Blimp has been first choice select regular first choice balloon.
3. If step 2 is not succesfull take a 6F guide extension and repeat sequence of step 1&2.
4. If step 3 is also not succesfull report how else succeeded (e.g. tonus, balloon rupture, carlino, rotablation, subintimal cross…) or not.

See also appendix I for a flow chart case situation A.

6.1.2 Case Situation B Small balloon catheter (≤ 1.5 (mm)) needed for procedure- no micro catheter used.

Case situation B is the circumstansis where a physician is in the stage of a procedure where he/ she would normally want to select a small balloon catheter ((≤ 1.5 (mm)) to cross an occluded or subtotlal stenotic segment of the coronary artery. When in such case the balloon catheter is not crossing the selection/ attempt with another balloon is one of the current common options as next step.

For the study the physician will go through following steps

1. select alternating in 50% of these cases his current first choice regular balloon (≤ 1.5 (mm) OD) and in the other 50% of cases the Blimp.
2. If first choice regular balloon does not cross select the Blimp and if the Blimp has been first choice select regular first choice balloon.
3. If step 2 is not succesfull take a 6F guide extension and repeat sequence of step 1&2.
4. If step 3 is also not succesfull report how else succeeded (e.g. tonus, balloon rupture, carlino, rotablation, subintimal cross…) or not.See also appendix I for a flow chart of case situation B.

6.1.3 Use of the Blimp during the study

The Blimp should be used conform its Instruction For Use (IFU). Following techniques can be attemted to cross the lesion.

1. Regular balloon crossing of lesion if no significant resistance is felt.
2. Application of distal force/ push to the tip of Blimp against the proximal cap of the occlusion/subtotal lesion for 5-10 seconds to allow cap penetration due to spring principle of Blimp shaft.
3. If no progressing in step 2 keep distal force/ push to the tip of the Blimp and inflate to 25-30 ATM to attempt wedging/ scoring of the proximal cap.
4. Repeat step 2&3 up to three times to see if proximal cap/ crossing progression is made.
5. If after multiple attemps of step 2&3 no progression is demonstrated it should be concluded that the Blimp was unsuccesfull in crossing.

6.1.4 Study population and number of subjects A total 128 patients which are being targeted for percutaneous coronary intervention are selected for this study. Pased on power calculations, 128 patiants are sufficient to demonstrate a statistical significant difference in outcome (P<0.05) with 80% power.

6.1.5 Inclusion/exclusion criteria Patients will be enrolled if they require percutaneous coronary intervention (PCI) procedure and

1. During the case a micro catheter is being used which is not able to cross after crossing of the guidewire (case situation A).
2. During the case a small balloon catheter (≤ 1.5 (mm) OD) is being used and is not able to cross the target lesion (case situation B) .

Patients which under normal conditions would be excluded for a PCI procedure by the hospital will be excluded from the study.

6.1.6 Rational and justification of chosen study design The Blimp is intended for balloon dilatation of a coronary artery subtotal lesion/occlusions.

Due to its

* very small profile
* high rated burst pressure and
* guidewire scoring element over the balloon

the device has several features which can improve the crossabiltiy and initial dilation of severe occluded vessels. The study has been designed such to investigate in an objective and controlled manner if the Blimp Scoring balloon is providing an improved procedural success rate in these matters.

ELIGIBILITY:
Inclusion Criteria:

* Severe coronary lesion where microcatheter or dilatation balloon does not cross

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-03-28 (Actual)

PRIMARY OUTCOMES:
Successful crossing through lesion and dilatation with BLIMP or low profile balloon | The primary outcome is a procedural assessment
  passing of BLIMP or low profile balloon through lesion. If device passess it will be determined a successful outcome, if it does not pass, an unsuccesful outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Johan Bennett, Leuven, Brabant
  - ZOL Genk, Genk

IPD SHARING:
Plan to Share IPD: No